CLINICAL TRIAL: NCT05078359
Title: Optimizing Positive Predicting Value of Prostate Magnetic Resonance Imaging: Retrospective Multi-institutional Study Using the PRostate Mri Outcome Database (PROMOD)
Brief Title: Optimizing Positive Predicting Value of Prostate MRI
Acronym: PROMOD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Ugo Giovanni Falagario, Urologist, Ospedali Riuniti di Foggia
Other Study IDs: OspedaliRFUrology01
Record Dates: First submitted 2021-09-22; First posted 2021-10-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate Magnetic resonance imaging; Prostate Biopsy; Biomarkers
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prostate Magnetic resonance Imaging — Magnetic resonance imaging (MRI) uses a magnetic field, radiofrequency pulses, and a computer to produce detailed pictures of the organ. Prostate MRI evaluate the presence and extent of prostate cancer and determine whether it has spread around the organ

SUMMARY:
The PROMOD study is an international multicenter retrospective Project. The aim is to create a comprehensive database that will include multiple heterogeneous cohorts in order to explore inter-center differences in the accuracy of Magnetic Resonance Imaging (MRI) in the diagnosis of prostate cancer and to define optimal strategies for the selection of men at risk of clinically significant prostate cancer who might benefit from biopsies.

DETAILED DESCRIPTION:
Background:

In the recent years Magnetic Resonance Imaging (MRI) of the prostate and targeted biopsy have been shown to substantially improve detection of International Society of Urological Pathology (ISUP) prostate cancer (PCa) Gleason Grade Group (GG) ≥ 2, clinically significant prostate cancer (csPCa). In fact, 2020 European Association of Urology (EAU) guidelines recommend performing MRI before prostate biopsy in men with prior negative prostate biopsy as well as in biopsy naive men with a clinical suspicion of PCa. If MRI is positive, a combination of targeted and systematic biopsy should be performed. If MRI is negative, biopsy could be omitted based on the clinical suspicion of PCa and a shared decision-making with the patient. Such approach binds the decision to perform biopsy to the clinical suspicion of PCa to be determined using MRI, risk calculators, and biomarkers. While several risk calculators and biomarkers have been developed and are currently under evaluation, the 'MRI pathway' is supported by level 1 evidence but seems to be limited by the low to moderate inter-reader and inter-center reproducibility and the low specificity/positive predictive value.

Additionally, several techniques for target prostate biopsies have been described but recent studies found no significant differences among various methods of MRI targeted biopsy for csPCa detection.

The aim of this international multicenter project is to create a comprehensive database including multiple heterogeneous cohorts in order to explore inter-center differences in the accuracy of MRI, and define optimal strategies for selection of men who might benefit from biopsies.

Objectives:

1. To investigate variables (such as lesion size, lesion location, number of biopsy cores per lesion) affecting the Positive predictive value (PPV) of prostate MRI on lesion level and patient level.
2. To explore inter-center differences in PPV of prostate MRI and possible reasons for such differences on lesion level and patient level
3. To evaluated combined use of MRI with prostate-specific antigen (PSA) and other clinical variables (such as age, race, history of prior negative prostate biopsy, use of 5-alpha-reductase inhibitor, family history of PCa/csPCa) in A. men with a clinical suspicion of PCa, B. men with diagnosed prostate cancer on active surveillance
4. To assess if there is an optimal cut-off of MRI suspicious scores and PSA density (PSAd) in each individual institution.

5) to assess the impact of patient selection on biopsy rate and number of men who could safely avoid biopsy despite MRI suspicious findings in per center and pooled data analyses

Outcome:

Histological evidence of Clinically significant Prostate Cancer (csPCa), defined as Gleason score 3+4 or higher.

Inclusion criteria:

* Patients who received prostate biopsy with a pre-biopsy MRI.
* Additional inclusion criteria will be project-specific.

Methods:

Deidentified data from each cohort will be collected in a RedCap HIPPA compliant Database. Each center is responsible for the deidentification of the shared spreadsheet. The data handling center will be the University of Foggia (Foggia, Italy) and datasets will not be imported until data transfer agreements are complete between the institution sending data and the data handling center.

Data analysis Retrospective analyses of multiple prospective single- and multi-institutional clinical trials and cohort studies. The analysis will be performed on per center level as well using pooled dataset and will include comparisons of MRI and clinical, blood variables in men who underwent A. target biopsy only, B. targeted and systematic biopsy, C. systematic biopsy only. Decision curve analysis will be performed to assess the biopsy strategy with the higher clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

Patients who received prostate biopsy with a pre biopsy MRI.

Exclusion Criteria:

Patients who underwent previous treatments for prostate cancer Patients who underwent post biopsy MRI

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing Prostate biopsy with a pre biopsy MRI and no previous treatmens
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinically significant prostate cancer detected at prostate biopsy | 3 to 5 weeks
  Number of patients with histological evidence of clinically significant prostate cancer (defined as histologic Gleason Score 3+4 or higher) in prostate biopsy cores.

CONTACTS AND LOCATIONS:
Locations (1):
- university ospital: Ospedali Riiuniti di Foggia, Foggia, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falagario UG, Lantz A, Jambor I, Busetto GM, Bettocchi C, Finati M, Ricapito A, Luzzago S, Ferro M, Musi G, Totaro A, Racioppi M, Carbonara U, Checcucci E, Manfredi M, D'Aietti D, Porcaro AB, Nordstrom T, Bjornebo L, Oderda M, Soria F, Taimen P, Aronen HJ, Perez IM, Ettala O, Marchioni M, Simone G, Ferriero M, Brassetti A, Napolitano L, Carmignani L, Signorini C, Conti A, Ludovico G, Scarcia M, Trombetta C, Claps F, Traunero F, Montanari E, Boeri L, Maggi M, Del Giudice F, Bove P, Forte V, Ficarra V, Rossanese M, Mucciardi G, Pagliarulo V, Tafuri A, Mirone V, Schips L, Antonelli A, Gontero P, Cormio L, Sciarra A, Porpiglia F, Bassi P, Ditonno P, Bostrom PJ, Messina E, Panebianco V, De Cobelli O, Carrieri G; PROMOD Study Group. Diagnosis of prostate cancer with magnetic resonance imaging in men treated with 5-alpha-reductase inhibitors. World J Urol. 2023 Nov;41(11):2967-2974. doi: 10.1007/s00345-023-04634-2. Epub 2023 Oct 3. PMID 37787941